CLINICAL TRIAL: NCT04875273
Title: Effects of Magnetic Tape on Perceived Spine Pain and Over Ankle Dorsiflexion in Patients With Low Back Pain: RCT
Brief Title: Effects of Magnetic Tape on Perceived Spine Pain and Over Ankle Dorsiflexion in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Selva (Other)
Responsible Party: Sponsor-Investigator, Francisco Selva, PhD physiotherapy, Clínica Dr. Francisco Selva
Organization: Clínica Dr. Francisco Selva (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2021-04-26; First posted 2021-05-06 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Back Pain
Keywords: pain; magnetic tape; algometer; low back pain; leg motion; Mobility; Range of motion
MeSH Terms: conditions — Back Pain; Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- Pre: pain assessment in the spinous processes of the spine with 1kg (No Intervention): press on the spinous processes with the algometer perpendicularly.
- Pre: pain assessment in the spinous processes of the spine with 2 kg (No Intervention): press on the spinous processes with the algometer perpendicularly.
- Pre: pain assessment in the spinous processes of the spine with 3 kg (No Intervention): press on the spinous processes with the algometer perpendicularly.
- Pre: pain assessment in the spinous processes of the spine with maximum pressure (No Intervention): press on the spinous processes with the algometer perpendicularly.
- Post Exp: pain assessment in the spinous processes of the spine with 1kg (Experimental): press on the spinous processes with the algometer perpendicularly.
  Interventions: Device: Magnetic Tape® aplicación
- Post Exp: pain assessment in the spinous processes of the spine with 2kg (Experimental): press on the spinous processes with the algometer perpendicularly.
  Interventions: Device: Magnetic Tape® aplicación
- Post Exp: pain assessment in the spinous processes of the spine with 3kg (Experimental): press on the spinous processes with the algometer perpendicularly.
  Interventions: Device: Magnetic Tape® aplicación
- Post Exp: pain assessment in the spinous processes of the spine with maximum pressure (Experimental): press on the spinous processes with the algometer perpendicularly.
  Interventions: Device: Magnetic Tape® aplicación
- Post Pla: pain assessment in the spinous processes of the spine with 1kg (Placebo Comparator): press on the spinous processes with the algometer perpendicularly.
  Interventions: Device: Kinesiology Tape application
- Post Pla: pain assessment in the spinous processes of the spine with 2kg (Placebo Comparator): press on the spinous processes with the algometer perpendicularly.
  Interventions: Device: Kinesiology Tape application
- Post Pla: pain assessment in the spinous processes of the spine with 3kg (Placebo Comparator): press on the spinous processes with the algometer perpendicularly.
  Interventions: Device: Kinesiology Tape application
- Post Pla: pain assessment in the spinous processes of the spine with maximum pressure (Placebo Comparator): press on the spinous processes with the algometer perpendicularly.
  Interventions: Device: Kinesiology Tape application
- Pre: Right Ankle Dorsiflexion (No Intervention): Range of motion in right ankle dorsiflexion is measured with LegMOtion®
- Post Pla: Right Ankle Dorsiflexion (Placebo Comparator): Range of motion in right ankle dorsiflexion is measured with LegMOtion®
  Interventions: Device: Kinesiology Tape application
- Post Exp: Right Ankle Dorsiflexion (Experimental): Range of motion in right ankle dorsiflexion is measured with LegMOtion®
  Interventions: Device: Magnetic Tape® aplicación
- Pre: Left Ankle Dorsiflexion (No Intervention): Range of motion in left ankle dorsiflexion is measured with LegMOtion®
- Post Pla: Left Ankle Dorsiflexion (Placebo Comparator): Range of motion in left ankle dorsiflexion is measured with LegMOtion®
  Interventions: Device: Kinesiology Tape application
- Post Exp: Left Ankle Dorsiflexion (Experimental): Range of motion in left ankle dorsiflexion is measured with LegMOtion®
  Interventions: Device: Magnetic Tape® aplicación

INTERVENTIONS:
Device: Magnetic Tape® aplicación — Magnetic tape® is applied without creating any tension on the paravertebral skin of the lumbar spine
  Arms: Post Exp: Left Ankle Dorsiflexion; Post Exp: Right Ankle Dorsiflexion; Post Exp: pain assessment in the spinous processes of the spine with 1kg; Post Exp: pain assessment in the spinous processes of the spine with 2kg; Post Exp: pain assessment in the spinous processes of the spine with 3kg; Post Exp: pain assessment in the spinous processes of the spine with maximum pressure
Device: Kinesiology Tape application — Kinesiology tape is applied without creating any tension on the paravertebral skin of the lumbar spine
  Arms: Post Pla: Left Ankle Dorsiflexion; Post Pla: Right Ankle Dorsiflexion; Post Pla: pain assessment in the spinous processes of the spine with 1kg; Post Pla: pain assessment in the spinous processes of the spine with 2kg; Post Pla: pain assessment in the spinous processes of the spine with 3kg; Post Pla: pain assessment in the spinous processes of the spine with maximum pressure

SUMMARY:
The tape will be applied on the lumbar area bilateralemten to the spine without creating any tension.

The possible variation in perceived pain in each spinous process is measured with the Wagner Force Dial-FDK 20 algometer.

The possible variation in the range of motion in ankle dorsiflexion is measured with LegMOtion® Therapeutic and Corrective Exercise Assessment System.

A kinesiology tape was used as a placebo tape and the magnetic tape was used in a randomized experimental way.

DETAILED DESCRIPTION:
A double-blind randomized clinical trial is designed where subjects with low back pain will be selected and blinded to recieve the Magnetic Tape® or placebo Tape. Likewise, the evaluator who puts the Magnetic Tape® does not know what material he is using, as it is supplied by another researcher.

The recommendations of the "Consolidated Standards of Reporting Trials" (CONSORT) will be followed. All participants will receive a participant information sheet and sign informed consent. Patients aged 18 to 65 years with low back pain will be recruited from different private clinics in the city of Valencia, Spain.

The hypothesis is that when Magnetic Tape® comes into contact with electromagnetic fields such as those generated by living beings, due to the movement of electrical charges (ions), as defined by Ampere's Law, the domains of the tape are oriented or aligned in parallel with the external magnetic field creating a magnetic flux with a north pole and a south pole. This generated field in turn produces a magnetic induction proportional to the variation of the magnetic flux, as defined by the Faraday Law.

This electric potential produces a redistribution of the electric charge (ions) generating a magnetic field due to the orientation of the tape domains, then exerting a force on the moving charges within the electrolyte.

Physiological, Lorentz's Law, regulating Magnetic Tape® aberrant electromagnetic fields.

After signing the informed consent and data protection, the groups with low back pain will be formed that will receive the application of both Magnetic Tape® and the intervention of a placebo tape. To avoid that the order of the intervention influences the results of the study, the subjects will be randomized into two different groups, Group A and Group B. Group A will receive Magnetic tape® and Group B will do the opposite. The next day the other tape will be applied.

The patient will be placed in the prone position and the spinous processes of L1 and L5 will be identified by marking them with a pen. Once L4 is located at the level of the iliac crests, the therapist will palpate the following spinous processes and will count down to the level of L1 and L5, and then mark it. The tapes are placed on the paravertebral muscles leaving the spinous processes uncovered by the tape.

Patients receive the two interventions on two different days and the tests serve as their own control. To avoid that the order of the intervention influences the results of the study, the subjects will be randomized into two different groups, Group A and Group B. Group A will be applied Magnetic tape® in their first visit and kinesiology tape or neuromuscular bandage in your next visit. Group B will do the opposite.

Before starting the research, a familiarization session will be held so that the assessments are consistent in terms of pain intensities using the VAS scale. To do this, an algometer will be pressed on the posterior deltoid at 2kg, 4kg and 6kg of pressure and later at 1kg, 2kg and 3kg of pressure, the EVA evaluations must coincide with the intensities of the pressures. Familiarization sessions will also be held so that the Lunge test are carried out properly and so that the results have the highest inter-observer reliability.

The perceived pain will be evaluated on two different days. The pain assessment in the spinous processes of the spine will be performed with the Wagner Force Dial-FDK 20 algometer, pressing at each level of the spine with 1kg, 2kg, 3kg and the maximum tolerable pressure separated by each measurement in time from at least one minute. During each press, the subject will rate perceived pain using the Visual Analog Pain Scale (VAS) while the subject is in the prone position.

Active joint ROM of both ankles is assessed by placing the patient in bipedestation. LegMOtion® will be used for to make measurements the Lunge test.

Neither application has to be painful.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with low back pain.
* Subjects aged 18-65 years.

Exclusion Criteria:

* Tape allergies
* Adhesive allergies
* Pregnant
* People with pacemakers
* People who have any contraindication of electromagnetic fields
* People with neurological diseases
* Taking any medication that may interact with magnetic fields.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-11 (Actual)

PRIMARY OUTCOMES:
Pressure | Changes in pain when applying pressure on the spinous processes, first evaluation before placing the tapes and immediately after placing the experimental tape and the placebo tape. It will wait at least one minute to repeat the test.
  pressure with 1kg, 2kg, 3kg and the maximum pressure in each spinous process.
Range of motion | Assessment System
  Maximum centimeters of ankle dorsiflexion measured with LegMOtion® Therapeutic and Corrective Exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Dr Francisco Selva, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No